CLINICAL TRIAL: NCT01819480
Title: A Single Arm Study of Efficacy and Functional Quality of Life in Patients Treated With Transoral Robotic Surgery for Oropharyngeal and Supraglottic Squamous Cell Carcinoma
Brief Title: Efficacy and Safety of TORS for SCCA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Katherine L Fedder (Other)
Responsible Party: Sponsor-Investigator, Katherine L Fedder, Principal Investigator, University of Virginia
Organization: University of Virginia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16376; 16376 (Other: University of Virginia IRB-HSR)
Record Dates: First submitted 2013-03-22; First posted 2013-03-27 (Estimated); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Oropharyngeal Squamous Cell Carcinoma; Supraglottic Squamous Cell Carcinoma
Keywords: Surgery; Robotic; Carcinoma; squamous cell of head and neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transoral robotic surgery (Experimental): Transoral robotic surgery
  Interventions: Procedure: Transoral robotic surgery

INTERVENTIONS:
Procedure: Transoral robotic surgery — Transoral robotic surgery using the daVinci robot to remove primary tumor

SUMMARY:
The purpose of this study is to learn more about the outcomes of treatment of throat and voice box cancers using transoral robotic surgery (TORS). TORS is a relatively new option involving the use of the da Vinci surgical robot to remove these cancers through the mouth.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female
* Diagnosis of either oropharyngeal or supraglottic squamous cell carcinoma

Exclusion Criteria:

* Metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2013-03; Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 3 years
  Duration of time from date of surgery to date of recurrence or death

SECONDARY OUTCOMES:
Disease specific survival | 3 years
  Duration of time from the date of surgery until death with disease present

OTHER OUTCOMES:
Overall survival | 3 years
  Measured from the date of surgery until date of death from any cause
Functional quality of life | 3 years
  Subject-reported functional outcome questionnaires will be used to quantify patient-reported speech and swallowing function
Incidence of adverse events | 3 years
  Adverse events occuring following the surgery will be reported and graded using CTCAE v4.0 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L Fedder, MD, Principal Investigator — University of Virginia School of Medicine
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States